CLINICAL TRIAL: NCT03620331
Title: Surgical Treatment of Peri-implantitis With and Without an Initial Non-surgical Approach: a Multi-center Randomized Clinical Trial
Brief Title: Surgical Treatment of Peri-implantitis With and Without an Initial Non-surgical Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Azienda Policlinico Umberto I (Other); University of Turin, Italy (Other); Osteology Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Peri-implantitis_ImmediateSurg
Record Dates: First submitted 2018-08-02; First posted 2018-08-08 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Peri-Implantitis
MeSH Terms: conditions — Peri-Implantitis | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non Surgical + Surgical (Active Comparator): Non surgical approach (NS) followed by surgical treatment (S) of peri-implantitis
  Interventions: Procedure: Surgery with a previous non-surgical approach
- Immediate Surgery (Experimental): Direct surgical approach (S), without a previous non surgical approach
  Interventions: Procedure: Surgery without a previous non-surgical approach

INTERVENTIONS:
Procedure: Surgery with a previous non-surgical approach — Non-surgical phase done prior to the surgical treatment of peri-implantitis
  Arms: Non Surgical + Surgical
Procedure: Surgery without a previous non-surgical approach — Non-surgical phase not done prior to the surgical treatment of peri-implantitis
  Arms: Immediate Surgery

SUMMARY:
Randomized, surgeon and outcome assessor blinded, multi-centric, superiority trial with two parallel groups and a 1:1 allocation ratio with the aim of comparing the surgical treatment of severe peri-implantitis with or without an initial non surgical approach.

ELIGIBILITY:
Inclusion Criteria:

Any patient having at least one implant affected by severe peri-implantitis, being at least 18 years old and able to sign an informed consent form will be potentially eligible for this trial.

Severe peri-implantitis will be defined as peri-implant probing pocket depth [PPD] ≥6 mm in at least 1 site of the implant, together with bleeding and/or suppuration on probing [BoP and/or SoP, respectively] and radiographically documented marginal bone loss/level ≥3 mm (Carcuac et al. 2016) on implants in function by at least 1 year. In case of absence of baseline radiographs, the reference point for baseline bone levels will be considered where bone was likely to be at implant placement.

Exclusion Criteria:

Patients fitting to all the inclusion criteria as above will be not included in the study if they appear to be unable to attend to the study-related procedures (including the follow-up visits) or if one or more of the following systemic or local exclusion criteria are found in the enrolment phase.

Systemic primary exclusion criteria:

* compromised general health which contraindicates the study procedures (ASA IV-VI patients);
* systemic diseases which could influence the outcome of the therapy (uncontrolled diabetes mellitus);
* pregnant or nursing women;
* chronic use of corticosteroids or NSAID or immune-modulator drugs (any type and any dose);
* patients who need use of medications affecting bone metabolism or peri-implant mucosa (bisphosphonates, any type and any dose).

Local primary exclusion criteria:

* history of peri-implantitis treatment on implants to be included in the study (included topical antibiotics);
* hopeless implants (e.g. mobility) to be included in the study.

Secondary exclusion criteria:

- uncompliant patients (poor oral hygiene 2 weeks after OHI).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Disease Resolution | 1 year post-surgery
Probing Pocket Depth changes | 1 year post-surgery
  Measured from the mucosal margin to the bottom of the probeable pocket.

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Sanz Alonso, Study Chair — Department of Periodontology, University Complutense Madrid, Spain; Luca Cordaro, Study Chair — Department of Periodontology and Prosthodontics, "Umberto I" Policlinic - "G. Eastman" Section; Mario Romandini, Study Director — Department of Periodontology, University Complutense Madrid, Spain
Locations (3):
- Italy (2):
  - Policlinico Umberto I - "G. Eastman" Section - Department of Periodontology, Roma
  - Department of Surgical Sciences, C.I.R. Dental School, University of Turin, Turin
- Department of Periodontology, University Complutense Madrid, Spain, Madrid, Spain

REFERENCES:
- [Derived] Romandini M, Lafori A, Pedrinaci I, Baima G, Ferrarotti F, Lima C, Paterno Holtzman L, Aimetti M, Cordaro L, Sanz M. Effect of sub-marginal instrumentation before surgical treatment of peri-implantitis: A multi-centre randomized clinical trial. J Clin Periodontol. 2022 Dec;49(12):1334-1345. doi: 10.1111/jcpe.13713. Epub 2022 Sep 9. PMID 36085409